CLINICAL TRIAL: NCT06045208
Title: Comparison of the Effects of Foot and Lower Extremity Strengthening Exercises in Adolescents With Pes Planovalgus
Brief Title: Foot and Lower Extremity Exercises in Adolescents With Pes Planovalgus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Halenur Evrendilek (Other)
Responsible Party: Sponsor-Investigator, Halenur Evrendilek, Research Assistant, Istanbul Kültür University
Organization: Istanbul Kültür University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/52
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Flat Foot
Keywords: exercise; foot posture; foot kinematic
MeSH Terms: conditions — Flatfoot; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foot Exercise Group (FEG) (Active Comparator)
  Interventions: Other: Foot exercise
- Lower Extremity Exercise Group (LEEG) (Active Comparator)
  Interventions: Other: Lower Extremity Exercise
- Control Group (CG) (No Intervention)

INTERVENTIONS:
Other: Foot exercise — This group will engage in an 8-week foot intrinsic strengthening training
  Arms: Foot Exercise Group (FEG)
Other: Lower Extremity Exercise — This group will engage in an 8-week lower extremity strengthening training
  Arms: Lower Extremity Exercise Group (LEEG)

SUMMARY:
The study aims to determine and compare the effects of 8-week intrinsic foot muscle-strengthening exercises and lower extremity strengthening exercises in adolescents with pes planovalgus.

ELIGIBILITY:
Inclusion Criteria:

* Age between the 12-18 years,
* Foot posture index-6 score > 6,
* Navicular drop test value > 1 cm,
* Body mass index between 18.5 - 25 kg/m2,
* Children with flexible pes planovalgus

Exclusion Criteria:

* Presence of any pathology that prevents participation in exercises
* Diagnosis of any neurological, psychological, or metabolic disease
* History of orthopedic surgery
* Use of insoles in the last 1 year
* Leg length discrepancy and scoliosis

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Foot posture assesment | Pre-intervention assesment and after 8-week
  Foot Posture Index 6 and navicular drop will be used for assesing the foot pronation.
Foot muscle strentgh assesment | Pre-intervention assesment and after 8-week
  Toe muscle strength will be assessed through the utilization of a handheld dynamometer.
Performance and dynamic balance assesment | Pre-intervention assesment and after 8-week
  Front jump test and star excursion balance test will be performed by participants.
3D gait analysis | Pre-intervention assesment and after 8-week
  The kinetic/kinematic analysis of the foot and the lower extremity will be conducted using a motion capture system, specifically employing the Oxford Foot Model and the Plug-in Gait Model.

SECONDARY OUTCOMES:
Functional assesment | Pre-intervention assesment and after 8-week
  The Oxford Ankle Foot Questionnaire for Children (OxAFQ-C) will be utilized for function-related aspect.
Quality of life assesment | Pre-intervention assesment and after 8-week
  Pediatric Quality of Life Inventory (PedsQL) will be utilized for the assessment of participants' quality of life status.

CONTACTS AND LOCATIONS:
Overall Officials: Halenur Evrendilek, MSc, PhD (c), Principal Investigator — Istanbul University - Cerrahpasa; Derya Çelik, Prof. Dr., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul Kultur University, Bahçelievler, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No